CLINICAL TRIAL: NCT01192672
Title: Use of Expressive Writing in Irritable Bowel Syndrome (IBS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: Takeda Pharmaceuticals North America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4764-8
Record Dates: First submitted 2010-08-12; First posted 2010-09-01 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Expressive Writing (Experimental): Subjects in the Intervention were instructed to write for 30-minute intervals for 4 consecutive days about their deepest thoughts and feelings related to their Irritable Bowel Syndrome.
  Interventions: Behavioral: Expressive Writing
- Control Writing (Active Comparator): The participants were instructed to write for 30-minute intervals for 4 consecutive days about all of the actions they performed that day for a 24 hour period. The subjects were asked not to write about their feelings or thoughts related to these actions.
  Interventions: Behavioral: Control Writing
- Usual Care (No Intervention): Subjects in this group did not receive an intervention. They filled out measures at baseline, 1 month, and 3 month follow-up time periods.

INTERVENTIONS:
Behavioral: Expressive Writing — Subjects in the Intervention were instructed to write for 30-minute intervals for 4 consecutive days about their deepest thoughts and feelings related to their Irritable Bowel Syndrome.
  Arms: Expressive Writing
Behavioral: Control Writing — Subjects were asked to write about the actions they performed during the last 24 hours. They were asked not to write about their feelings or thoughts related to these actions.
  Arms: Control Writing

SUMMARY:
The purpose of this study is to test whether disease-related expressive writing is effective in the treatment of Irritable Bowel Syndrome (IBS).

DETAILED DESCRIPTION:
Expressive writing involves writing about traumatic, stressful or emotional events. Expressive writing, for as little as 3-5 sessions of 20 minutes, has been found to improve both physical and psychological health based on health outcome measures such as number of doctor's visits and hospital days, blood pressure control, lung and immune function, and pain. Given its simplicity, and obvious advantages in terms of cost efficiency, expressive writing appears to have great potential as a therapeutic tool or as a means of self-help, either alone or as an adjunct to traditional therapies. This modality has not been studied in irritable bowel syndrome (IBS), a common gastrointestinal condition, which is lacking well-defined etiology or treatments and is best understood in a biopsychosocial context.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Irritable Bowel syndrome

Exclusion Criteria:

* Non-English Speakers

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2008-09 (Actual); Primary Completion 2010-09 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
IBS-Specific Quality of Life (IBS-QOL) | 3 months
  IBSQOL is a measure of IBS - specific quality of life.

SECONDARY OUTCOMES:
CT3 | 3 months
  Measure of health-related cognition (catastrophizing or maladaptive coping,and patients' perceived ability to control symptoms)
Health care Utilization (HCU) | 3 months
  HCU is a measure of frequency and type of health care received for IBS
IBSSS | 3 months
  IBSSS provides a disease severity measure
Demographics (DEM-MED) | Baseline
  Demographic information
Cognitive Scale for Functional Bowel Disorders (CGFBD) | 3 months
  Measure of IBS related cognitions.
Writing Evaluation Questionnaire (WEQ) | 3 months
  The WEQ measure obtains subjects' reflections about their writing experience.

CONTACTS AND LOCATIONS:
Overall Officials: Albena Halpert, MD, Principal Investigator — Boston University

IPD SHARING:
Plan to Share IPD: No